CLINICAL TRIAL: NCT00539591
Title: Phase II Study Incorporating Pegylated Interferon In the Treatment For Children With High-Risk Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEL06; NCI-2011-01192 (Registry Identifier: NCI Clinical Trials Registration Program ID)
Record Dates: First submitted 2007-10-02; First posted 2007-10-04 (Estimated); Results first posted 2014-02-27 (Estimated); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Malignant Melanoma
Keywords: Cutaneous Melanoma
MeSH Terms: conditions — Melanoma | interventions — peginterferon alfa-2b; Temozolomide; Introns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Temozolomide/peginterferon alfa-2b (Experimental): Stratum B: Resected Stage IIIC, unresectable Stage III, Stage IV, and recurrent patients
  Stratum B is divided into 2 groups based on the presence (Stratum B1) or absence (Stratum B2) of measurable disease. Subjects will receive 8 weekly doses of peginterferon alfa-2b 0.5 mcg/kg/dose subcutaneously (SQ) in combination with temozolomide 75mg/m2/dose by mouth (PO) daily for 6 weeks followed by 2 week break. The duration of each treatment course will be 8 weeks. Strata B2 (no measurable disease) will proceed with 7 courses as outlined.
  Interventions: Drug: Peginterferon alfa-2b; Drug: Temozolomide
- Peginterferon alfa-2b/non-pegylated interferon alfa-2b (Experimental): Stratum A: Resected Stages IIC, IIIA, and IIIB patients will receive recombinant interferon alfa-2b 20 million units/m2/day intravenously (IV) 5 consecutive days per week for 4 weeks followed by peginterferon alfa-2b 1mcg/kg subcutaneously (SQ) once a week for 48 weeks.
  Interventions: Drug: Peginterferon alfa-2b; Drug: Temozolomide; Drug: Recombinant interferon alfa-2b

INTERVENTIONS:
Drug: Peginterferon alfa-2b — Given either IV or SQ. Therapeutic drug class: interferon.
  Other Names: PEG-Intron(R); pegylated interferon alfa-2b
Drug: Temozolomide — Given PO. Therapeutic drug class: antineoplastic agent.
  Other Names: Temodar(R), SCH 52365
Drug: Recombinant interferon alfa-2b — Given IV. Therapeutic drug classes: antineoplastic agent, immunomodulatory agent, interferon
  Other Names: Intron®; non-pegylated interferon alfa-2b
  Arms: Peginterferon alfa-2b/non-pegylated interferon alfa-2b

SUMMARY:
The main goal of this study is to estimate the tumor response rate of temozolomide administered in combination with peginterferon alfa-2b to pediatric patients with unresectable Stage III, metastatic, or recurrent cutaneous melanoma.

DETAILED DESCRIPTION:
This study is for children with malignant melanoma and high risk features (at high risk of melanoma returning or spreading to other parts of the body) or who have recurrent disease. The study has two treatment groups based on the stage of the disease. Patients with stage IIC, IIIA or IIIB melanoma whose tumors have been removed by surgery will be treated in study group A. These patients will receive 4 weeks of high dose interferon alfa-2b followed by 48 weeks of peginterferon. Patients with stage IIIC or IV melanoma, stage III melanoma that could not be removed by surgery and those with recurrent disease will be treated in study group B. These patients will receive peginterferon alfa-2b and temozolomide.

Stratum A: Resected Stages IIC, IIIA, and IIIB patients

Induction therapy (weeks 1-4): Subjects will receive recombinant interferon alfa-2b 20 million units/m2 per day intravenously over 20-30 minutes on 5 consecutive days per week for 4 weeks. Subjects will receive peginterferon alfa-2b 1 mcg/kg/week subcutaneously for a total of 48 weeks.

Stratum B: Resected Stage IIIC, unresectable Stage III, Stage IV, and recurrent patients

Stratum B is divided into 2 groups based on the presence (Stratum B1) or absence (Stratum B2) of measurable disease. Subjects will receive 8 weekly doses of peginterferon alfa-2b 0.5 mcg/kg/dose subcutaneously in combination with temozolomide 75mg/m2/dose by mouth daily for 6 weeks followed by 2 week break. The duration of each treatment course will be 8 weeks. Strata B2 (no measurable disease) will proceed with 7 courses as outlined.

Surgery interventions -Associated with both Strata A and B Surgery description: All subjects with initial presentation of melanoma (T1-4) will be treated with primary wide local excision with a minimum of 1cm margin (if anatomically feasible) surrounding the primary lesion or biopsy scar. For lesions with Breslow's thickness of > 1mm or <or= with ulceration or Clark's level IV/V, a 2 cm margin is preferred when anatomically feasible. Subjects with sentinel lymph node(s) positive for disease, will undergo complete lymph node dissection of the involved nodal basin.

Additional objectives include:

* To assess the safety of temozolomide administered in combination with peginterferon α-2b to pediatric patients with resected AJCC Stage IIIC, unresectable Stage III, metastatic, or recurrent cutaneous melanoma (Stratum B).
* To study the feasibility and safety of administering peginterferon α-2b weekly for 48 weeks following an initial induction phase with intravenous high dose interferon α-2b for 4 weeks to pediatric patients with resected thick melanomas (> 4mm) with ulcerations (AJCC Stage IIC) and resected melanomas with regional lymph node metastases (AJCC Stage IIIA and IIIB) (Stratum A).

ELIGIBILITY:
Inclusion Criteria:

* AJCC stage IIC, III, IV or recurrent cutaneous melanoma
* Adequate bone marrow function
* Age less than or equal to 21 years of age at diagnosis
* Adequate liver and kidney function

Exclusion Criteria:

* Prior Therapy with dacarbazine or temozolomide
* Patients who have uncontrolled infection
* Patients with autoimmune hepatitis
* Patients who have a history of depression or other psychiatric diseases requiring hospitalization
* Patients taking systemic corticosteroids including oral steroids (i.e. prednisone, dexamethasone) or topical steroid creams/ointments. Steroid containing inhalers, steroid replacement for adrenal insufficiency and steroid premedication for prevention of transfusion or imaging contrast-agent related allergic reaction will be permitted.
* Patients with hypersensitivity reaction to non-pegylated interferon α-2b are not eligible for study
* Patients with diabetes mellitus not adequately controlled with medication
* Patients with hypo- or hyperthyroidism not adequately controlled with medication.
* Patients with a history of myocardial infarction, severe or unstable angina, or severe peripheral vascular disease.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2008-05-09 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2026-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Pappo, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (3):
- United States (3):
  - Rady Children's Hospital, San Diego, California
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Cancer Hospital at UT M.D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 29 patients were enrolled between May 9, 2008 and August 22, 2012. Of the 29 participants, 21 were enrolled at St. Jude Children's Research Hospital (SJCRH), 7 at MD Anderson, and 1 at Rady Children's Hospital. Twenty-three participants met stratum A eligibility, 2 met stratum B1 eligibility and 4 met stratum B2 eligibility.
Groups:
- Peginterferon ɑ-2b/Non-pegylated Interferon ɑ-2b: Stratum A: American Joint Committee on Cancer (AJCC) resected Stages IIC, IIIA, and IIIB
  Participants received recombinant interferon ɑ-2b 20 million units/m^2/day intravenously 5 consecutive days per week for 4 weeks followed by peginterferon ɑ-2b 1 mcg/kg subcutaneously once a week for 48 weeks.
- Temozolomide/Peginterferon ɑ-2b With Measureable Disease: Stratum B1: American Joint Committee on Cancer (AJCC) resected Stage IIIC, unresectable Stage III, Stage IV, and recurrent participants with measurable disease
  Participants received 8 weekly doses of peginterferon ɑ-2b 0.5 mcg/kg/dose subcutaneously in combination with temozolomide 75 mg/m^2/dose by mouth daily for 6 weeks followed by 2 week break. The duration of each treatment course was 8 weeks.
- Temozolomide/Peginterferon ɑ-2b Without Measureable Disease: Stratum B2: American Joint Committee on Cancer (AJCC) resected Stage IIIC, unresectable Stage III, Stage IV, and recurrent participants without measurable disease
  Participants received 8 weekly doses of peginterferon ɑ-2b 0.5 mcg/kg/dose subcutaneously in combination with temozolomide 75 mg/m^2/dose by mouth daily for 6 weeks followed by 2 week break. The duration of each treatment course was 8 weeks. Stratum B2 (no measurable disease) proceeded with 7 courses as outlined.
Period: Overall Study
Arm/Group | Peginterferon ɑ-2b/Non-pegylated Interferon ɑ-2b | Temozolomide/Peginterferon ɑ-2b With Measureable Disease | Temozolomide/Peginterferon ɑ-2b Without Measureable Disease
Started | 23 | 2 | 4
Completed | 18 | 0 | 1
Not Completed | 5 | 2 | 3
Not completed — Toxicity | 3 | 0 | 0
Not completed — Disease progression | 2 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peginterferon ɑ-2b/Non-pegylated Interferon ɑ-2b | Temozolomide/Peginterferon ɑ-2b With Measureable Disease | Temozolomide/Peginterferon ɑ-2b Without Measureable Disease | Total
Number analyzed (Participants) | 23 | 2 | 4 | 29
Age, Continuous [Median (Full Range); unit: years] | 10.3 (2.4) [2.4 to 20.0] | 11.9 (3.96) [3.96 to 19.89] | 18.4 (3.6) [3.6 to 22.1] | 10.77 (2.4) [2.4 to 22.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 0 | 1 | 16
  Male | 8 | 2 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Rate
Description: Tumor response rate of stratum B1 participants was evaluated after 1 treatment course of temozolomide plus peginterferon ɑ-2b. Complete response (CR) and partial response (PR) confirmed with repeated scan at least 4 weeks apart following completion of course 1 therapy. CR defined as disappearance of all target and non-target lesions with no new lesions detected. If available, no disease must be detected by immunocytology or serum tumor markers. PR defined as at least 30% decrease in disease measurement compared to disease measurement at study entry with no new lesions detected. Progressive disease (PD) defined as at least 20% increase in the disease measurement compared to the smallest disease measurement recorded since start of treatment, or appearance of one or more new lesions. Stable disease defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD compared to smallest disease measurement since start of treatment.
Time Frame: 8 weeks
Measure: Number; unit: participants
Groups:
- Stratum B1: Stratum B: American Joint Committee on Cancer (AJCC) resected Stage IIIC, unresectable Stage III, Stage IV, and recurrent participants, divided into 2 groups based on presence (B1) or absence (B2) of measurable disease
  Stratum B1 had presence of measurable disease. Participants received 8 weekly doses of peginterferon ɑ-2b 0.5 mcg/kg/dose subcutaneously in combination with temozolomide 75 mg/m^2/dose by mouth daily for 6 weeks followed by 2 week break. The duration of each treatment course was 8 weeks.
  Interventions: Temozolomide, peginterferon ɑ-2b
Arm/Group | Stratum B1
Number analyzed (Participants) | 2
participants
  Progressive Disease | 2
  Clinical Remission | 0

2. Primary Outcome: Number of Patients Who Experience Toxicity at or Above the Target Toxicity for Strata B1 and B2
Description: The objective was to assess the safety of temozolomide administered in combination with peginterferon a-2b in Stratum B participants.
  Accrual was suspended any time during therapy if 2 or more of 6, 4 or more of 12, 6 or more of 18, 8 or more of 24, 10 or more of 30 participants experienced target toxicity defined as:
  * Grade 4 non-hematologic (non-hem) toxicity that does not resolve to ≤grade 1 within 2 weeks from the time next dose is due and is determined to be probably or definitely related to protocol therapy
  * Grade 4 non-hem toxicity that is NOT constitutional symptoms (fever, chills, fatigue and/or pain)
  * Grade 3 elevations in creatinine or BUN that are determined to be probably or definitely related to protocol therapy
  * Grade 4 cardiopulmonary toxicity that is determined to be probably or definitely related to protocol therapy
  * Grade 4 mood alteration (suicidal ideation; danger to self or others)
Time Frame: 52 weeks
Population: This toxicity report was based on intention to treat population (ITT), all patients enrolled were included. The study did not meet its accrual goals within the planned timeframe due to slow accrual.
Measure: Number; unit: participants
Arm/Group | Temozolomide/Peginterferon ɑ-2b With Measureable Disease | Temozolomide/Peginterferon ɑ-2b Without Measureable Disease
Number analyzed (Participants) | 2 | 4
participants | 0 | 0

3. Primary Outcome: Number of Patients Who Experience Toxicity at or Above the Target Toxicity for Stratum A Patients
Description: The objective was to study the feasibility and safety of administering peginterferon a-2b weekly for 48 weeks following the initial induction phase to Stratum A participants.
  Accrual was suspended during the 48-week course if 2 or more of 6, 4 or more of 12, 6 or more of 18, 8 or more of 24, 10 or more of 30 participants experienced target toxicity defined as:
  * Grade 4 non-hematologic (non-hem) toxicity that does not resolve to ≤grade 1 within 2 weeks from the time next dose is due and is determined to be probably or definitely related to protocol therapy
  * Grade 4 non-hem toxicity that is NOT constitutional symptoms (fever, chills, fatigue and/or pain)
  * Grade 3 elevations in creatinine or BUN that are determined to be probably or definitely related to protocol therapy
  * Grade 4 cardiopulmonary toxicity that is determined to be probably or definitely related to protocol therapy
  * Grade 4 mood alteration (suicidal ideation; danger to self or others)
Time Frame: 52 weeks
Population: Number of participants for the analysis was based on the intent to treat population, all patients enrolled were included. Participants were enrolled on Stratum A until the accrual goals were met on Stratum B.
Measure: Number; unit: participants
Arm/Group | Peginterferon ɑ-2b/Non-pegylated Interferon ɑ-2b
Number analyzed (Participants) | 23
participants
  Grade 4 non-hem toxicity | 2
  Grade 4 non-hem/NOT constitutional | 0
  Grade 3 elevations in creatinine or BUN | 0
  Grade 4 cardiopulmonary toxicity | 0
  Grade 4 mood alteration | 1

4. Primary Outcome: Probability of Event-free Survival (EFS) of Stratum A Participants
Description: The probability of EFS was estimated as time to first event (relapse, death or second malignancy). As of April 2016, 21 out of 23 participants had no events. The EFS rate was estimated by Kaplan-Meier method.
Time Frame: 3 years from diagnosis
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Peginterferon ɑ-2b/Non-pegylated Interferon ɑ-2b
Number analyzed (Participants) | 23
probability | 0.913 [0.79 to 1.00]

5. Other Pre Specified Outcome: Median Steady State Trough Concentration of Pegylated Interferon ɑ-2B
Description: The pharmacokinetic (PK) analysis of pegylated ɑ-2b included only patients within Stratum A who had PK studies performed.
  Samples were analyzed for pegylated interferon ɑ-2b concentrations by using the VeriKine Human Interferon Alpha ELISA Kit following the manufacturer's instructions, and concentration-time data were analyzed by nonlinear-mixed effects modeling as implemented in NONMEM.
Time Frame: Before first dose, and 24, 96 and 168 hours after dose during weeks 5 and 28
Population: Only one patient had evaluable data in Stratum B and is not included in the final analysis, because data from more than one patient are required for nonlinear-mixed effects modeling.
Measure: Median (Full Range); unit: pcg/ml
Groups:
- Peginterferon ɑ-2b/Non-Pegylated Interferon ɑ-2b: Stratum A participants who received pegylated interferon ɑ-2b and had pharmacokinetic studies performed are included.
Arm/Group | Peginterferon ɑ-2b/Non-Pegylated Interferon ɑ-2b
Number analyzed (Participants) | 16
pcg/ml | 52.8 [13.8 to 152.4]

6. Other Pre Specified Outcome: Area Under the Curve (AUC) of Pegylated Interferon ɑ-2B
Description: Pharmacokinetic (PK) analysis of pegylated ɑ-2b included only Stratum A patients who had PK studies performed.
  Samples were analyzed for pegylated interferon ɑ-2b concentrations by using the VeriKine Human Interferon Alpha ELISA Kit following the manufacturer's instructions, and concentration-time data were analyzed by nonlinear-mixed effects modeling as implemented in NONMEM. AUC is given as Time 0 through infinity.
Time Frame: Before first dose, and 24, 96 and 168 hours after dose during weeks 5 and 28
Population: Only one Stratum B patient had evaluable data and is not included in final analysis, because data from more than one patient are required for nonlinear-mixed effects modeling. Two patients in Week 5 and three in Week 28 were excluded due to inadequate sampling to characterize an AUC value.
Measure: Median (Full Range); unit: pcg * hr/ml
Groups:
- Week 5 - First Dose: Stratum A participants who received pegylated interferon ɑ-2b and had pharmacokinetic studies performed are included.
- Week 28 - Steady State: Stratum A participants who received pegylated interferon ɑ-2b and had pharmacokinetic studies performed.
Arm/Group | Week 5 - First Dose | Week 28 - Steady State
Number analyzed (Participants) | 7 | 6
pcg * hr/ml | 50556 [36166 to 58980] | 48480 [34024 to 59857]

7. Other Pre Specified Outcome: ɑ Half Life of Pegylated Interferon ɑ-2B
Description: Pharmacokinetic (PK) analysis of pegylated ɑ-2b included only Stratum A patients who had PK studies performed.
  Samples were analyzed for pegylated interferon ɑ-2b concentrations by using the VeriKine Human Interferon Alpha ELISA Kit following the manufacturer's instructions, and concentration-time data were analyzed by nonlinear-mixed effects modeling as implemented in NONMEM.
Time Frame: Before first dose, and 24, 96 and 168 hours after dose during weeks 5 and 28
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | Peginterferon ɑ-2b/Non-Pegylated Interferon ɑ-2b
Number analyzed (Participants) | 9
hours | 24.8 [16.6 to 40.6]

8. Other Pre Specified Outcome: Volume of Central Compartment (Vc) of Pegylated Interferon ɑ-2B
Description: as for outcome 7
Time Frame: Before first dose, and 24, 96 and 168 hours after dose during weeks 5 and 28
Population: Only one Stratum B patient had evaluable data and is not included in final analysis, because data from more than one patient are required for nonlinear-mixed effects modeling due to differences in clinical variables. Two patients in Week 5 and three in Week 28 were excluded due to inadequate sampling to characterize an AUC value.
Measure: Median (Full Range); unit: ml/kg
Arm/Group | Peginterferon ɑ-2b/Non-Pegylated Interferon ɑ-2b
Number analyzed (Participants) | 9
ml/kg | 772 [594 to 1410]

9. Other Pre Specified Outcome: Apparent Clearance (CL) of Pegylated Interferon ɑ-2B
Description: as for outcome 7
Time Frame: Before first dose, and 24, 96 and 168 hours after dose during weeks 5 and 28
Population: Only one Stratum B patient had evaluable data and is not included in final analysis due to differences in clinical variables, because data from more than one patient are required for nonlinear-mixed effects modeling. Two patients in Week 5 and three in Week 28 were excluded due to inadequate sampling to characterize an AUC value.
Measure: Median (Full Range); unit: ml/hr/kg
Arm/Group | Peginterferon ɑ-2b/Non-Pegylated Interferon ɑ-2b
Number analyzed (Participants) | 9
ml/hr/kg | 19.8 [16.7 to 31.4]

10. Other Pre Specified Outcome: Area Under the Curve (AUC) of Interferon ɑ-2b
Description: Samples were analyzed for interferon ɑ-2b concentrations by using the VeriKine Human Interferon Alpha ELISA Kit following the manufacturer's instructions, and concentration-time data were analyzed by nonlinear-mixed effects modeling as implemented in NONMEM. AUC is given as Time 0 to infinity.
Time Frame: Before first dose, and 1, 2, 4, 6, 8, 12, and 24 hours postinfusion
Population: The pharmacokinetic(PK) analysis of pegylated ɑ-2b included only patients within Stratum A who had PK studies performed. Only one patient had evaluable data in Stratum B and is not included in the final analysis due to differences in clinical variables.
Measure: Median (Full Range); unit: pcg * hr/ml
Groups:
- Peginterferon ɑ-2b/Non-Pegylated Interferon ɑ-2b: Stratum A participants who received interferon ɑ-2b and had pharmacokinetic studies performed are included.
Arm/Group | Peginterferon ɑ-2b/Non-Pegylated Interferon ɑ-2b
Number analyzed (Participants) | 16
pcg * hr/ml | 5026 [2642 to 10270]

11. Other Pre Specified Outcome: Half-Life of Interferon ɑ-2b
Description: Samples were analyzed for interferon ɑ-2b concentrations by using the VeriKine Human Interferon Alpha ELISA Kit following the manufacturer's instructions, and concentration-time data were analyzed by nonlinear-mixed effects modeling as implemented in NONMEM.
Time Frame: Before first dose, and 1, 2, 4, 6, 8, 12, and 24 hours postinfusion
Population: The pharmacokinetic (PK) analysis of pegylated ɑ-2b included only patients within Stratum A who had PK studies performed. Only one patient had evaluable data in Stratum B and is not included in the final analysis due to differences in clinical variables.
Measure: Median (Full Range); unit: hours
Arm/Group | Peginterferon ɑ-2b/Non-Pegylated Interferon ɑ-2b
Number analyzed (Participants) | 16
hours
  ɑ half-life | 0.7 [0.4 to 1.4]
  ß half-life | 14.7 [12.5 to 28.2]

12. Other Pre Specified Outcome: Volume of Central Compartment (Vc) of Interferon ɑ-2b
Description: as for outcome 11
Time Frame: Before first dose, and 1, 2, 4, 6, 8, 12, and 24 hours postinfusion
Population: as for outcome 11
Measure: Median (Full Range); unit: l/m^2
Groups:
- Interferon ɑ-2b: Participants who received interferon ɑ-2b and had pharmacokinetic studies performed are included.
Arm/Group | Interferon ɑ-2b
Number analyzed (Participants) | 16
l/m^2 | 25.1 [13.9 to 49.2]

13. Other Pre Specified Outcome: Systemic Clearance (CL) of Interferon ɑ-2B
Description: as for outcome 11
Time Frame: Before first dose, and 1, 2, 4, 6, 8, 12, and 24 hours postinfusion
Population: as for outcome 11
Measure: Median (Full Range); unit: l/hr/m^2
Arm/Group | Interferon ɑ-2b
Number analyzed (Participants) | 16
l/hr/m^2 | 15.3 [7.5 to 29.1]

14. Other Pre Specified Outcome: Mean Total PedsQL 4.0 Scores for Child Quality of Life (QoL) Assessments (Stratum A)
Description: QoL assessments were completed using Pediatrics Quality of Life Inventory (PedsQL v4.0). Scale range is 0-100 with higher scores reflecting better quality of life. PedsQL 4.0 healthy sample normative mean ± SD for child report = 83.0 ± 14.8.
Time Frame: Pretherapy; Weeks 2, 4, 8, 12, and 24; and End of therapy at 6 months and 12 months post
Population: This QOL analysis included patients only within Stratum A.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pretherapy: QoL assessment completed before start of therapy.
- Week 2: QoL assessment completed at Week 2.
- Week 4: QoL assessment completed at Week 4.
- Week 8: QoL assessment completed at Week 8.
- Week 12: QoL assessment completed at Week 12.
- Week 24: QoL assessment completed at Week 24.
- End of Therapy: QoL assessment completed at end of therapy.
- 6 Months After End of Therapy: QoL assessment completed 6 months after end of therapy.
- 12 Months After End of Therapy: QoL assessment completed 12 months after end of therapy.
Arm/Group | Pretherapy | Week 2 | Week 4 | Week 8 | Week 12 | Week 24 | End of Therapy | 6 Months After End of Therapy | 12 Months After End of Therapy
Number analyzed (Participants) | 15 | 15 | 17 | 14 | 14 | 17 | 15 | 13 | 15
units on a scale | 75.5 (18.4) | 71.6 (18.7) | 77.2 (16.3) | 79.3 (17.4) | 77.8 (20.6) | 80.6 (15.6) | 80.4 (16.1) | 87.5 (12.5) | 91.0 (7.1)

15. Other Pre Specified Outcome: Mean Total PedsQL 4.0 Scores for Child Quality of Life (QoL) Assessments (Stratum B)
Description: as for outcome 14
Time Frame: Pretherapy; Weeks 2, 4, 8, 12, and 24; and End of therapy at 6 months and 12 months post
Population: Only one patient had evaluable data in Stratum B. The raw score, rather than the mean +/- SD, is presented. Data was not collected at Week 24, and the patient was taken off study prior to 6 months after end of therapy.
Measure: Number; unit: units on a scale
Arm/Group | Pretherapy | Week 2 | Week 4 | Week 8 | Week 12 | Week 24 | End of Therapy | 6 Months After End of Therapy | 12 Months After End of Therapy
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0
units on a scale | 90.3 | 93.1 | 72.8 | 79.2 | 68.1 |  | 65.6 |  |

16. Other Pre Specified Outcome: Mean Total PedsQL 4.0 Scores for Parent Quality of Life Assessments (Stratum A)
Description: QoL assessments were completed using Pediatrics Quality of Live Inventory (PedsQL v4.0). Scale range is 0-100 with higher scores reflecting better quality of life. PedsQL 4.0 healthy sample normative mean ± SD for parent report = 87.6 ± 12.3.
Time Frame: Pretherapy; Weeks 2, 4, 8, 12, and 24; and End of therapy at 6 months and 12 months post
Population: This QOL analysis included patients only within Stratum A.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pretherapy | Week 2 | Week 4 | Week 8 | Week 12 | Week 24 | End of Therapy | 6 Months After End of Therapy | 12 Months After End of Therapy
Number analyzed (Participants) | 16 | 15 | 17 | 13 | 16 | 17 | 15 | 15 | 15
units on a scale | 70.3 (19.1) | 71.8 (16.4) | 74.4 (17.9) | 79.1 (16.6) | 79.0 (19.0) | 82.2 (14.5) | 87.5 (15.3) | 86.0 (17.6) | 87.3 (17.5)

17. Other Pre Specified Outcome: Mean Total PedsQL 4.0 Scores for Parent Quality of Life Assessments (Stratum B)
Description: as for outcome 16
Time Frame: Pretherapy; Weeks 2, 4, 8, 12, and 24; and End of therapy at 6 months and 12 months post
Population: Only one patient had evaluable data in Stratum B. The raw score, rather than the mean +/- SD, is presented. Data was not collected after Week 4.
Measure: Number; unit: units on a scale
Arm/Group | Pretherapy | Week 2 | Week 4 | Week 8 | Week 12 | Week 24 | End of Therapy | 6 Months After End of Therapy | 12 Months After End of Therapy
Number analyzed (Participants) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
units on a scale | 77.6 | 72.2 | 89.1 |  |  |  |  |  |

18. Other Pre Specified Outcome: Mean Total PedsQL 3.0 Scores for Child Cancer Quality of Life (QoL) Assessments (Stratum A)
Description: QoL assessments were completed using Pediatrics Cancer Quality of Life Inventory (PedsQL v3.0). Scale range is 0-100 with higher scores reflecting better quality of life.
Time Frame: Weeks 2, 4, 8, 12, and 24; and End of therapy at 6 months and 12 months post
Population: PedsQL v3.0 was not completed pretherapy. This QOL analysis included patients only within Stratum A.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Week 2 | Week 4 | Week 8 | Week 12 | Week 24 | End of Therapy | 6 Months After End of Therapy | 12 Months After End of Therapy
Number analyzed (Participants) | 17 | 19 | 17 | 17 | 16 | 17 | 15 | 15
units on a scale | 71.1 (17.2) | 76.1 (15.4) | 79.2 (19.2) | 78.5 (14.7) | 77.1 (16.0) | 77.0 (16.5) | 83.7 (18.0) | 85.4 (8.9)

19. Other Pre Specified Outcome: Mean Total PedsQL 3.0 Scores for Child Cancer Quality of Life (QoL) Assessments (Stratum B)
Description: as for outcome 18
Time Frame: Weeks 2, 4, 8, 12, and 24; and End of therapy at 6 months and 12 months post
Population: PedsQL v3.0 was not completed pretherapy. Only one patient had evaluable data in Stratum B. The raw score, rather than the mean +/- SD, is presented. Data was not collected at Week 24, and the patient was taken off study prior to 6 months after end of therapy.
Measure: Number; unit: units on a scale
Arm/Group | Week 2 | Week 4 | Week 8 | Week 12 | Week 24 | End of Therapy | 6 Months After End of Therapy | 12 Months After End of Therapy
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0
units on a scale | 92.8 | 90.1 | 93.2 | 79.6 |  | 67.4 |  |

20. Other Pre Specified Outcome: Mean Total PedsQL 3.0 Scores for Parent Cancer Quality of Life (QoL) Assessments (Stratum A)
Description: as for outcome 18
Time Frame: Weeks 2, 4, 8, 12, and 24; and End of therapy at 6 months and 12 months post
Population: PedsQL v3.0 was not completed pretherapy. This QOL analysis included patients only within Stratum A.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Week 2 | Week 4 | Week 8 | Week 12 | Week 24 | End of Therapy | 6 Months After End of Therapy | 12 Months After End of Therapy
Number analyzed (Participants) | 19 | 19 | 17 | 18 | 16 | 16 | 15 | 15
units on a scale | 73.2 (13.9) | 75.1 (15.2) | 81.4 (11.6) | 78.7 (17.7) | 81.6 (17.1) | 85.6 (13.8) | 85.0 (11.5) | 89.1 (11.6)

21. Other Pre Specified Outcome: Mean Total PedsQL 3.0 Scores for Parent Cancer Quality of Life (QoL) Assessments (Stratum B)
Description: as for outcome 18
Time Frame: Weeks 2, 4, 8, 12, and 24; and End of therapy at 6 months and 12 months post
Population: PedsQL v3.0 was not completed pretherapy. Only one patient had evaluable data in Stratum B. The raw score, rather than the mean +/- SD, is presented. Data was not collected after Week 4.
Measure: Number; unit: units on a scale
Arm/Group | Week 2 | Week 4 | Week 8 | Week 12 | Week 24 | End of Therapy | 6 Months After End of Therapy | 12 Months After End of Therapy
Number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
units on a scale | 67.7 | 71.4 |  |  |  |  |  |

22. Other Pre Specified Outcome: BASC-2 Psychological Assessment (Stratum A)
Description: The Behavioral Assessment System for Children, 2nd Edition (BASC-2) was administered to parents, assessing for any effects on behavior or mood in children undergoing study therapy. The behavior system index (BSI) T-score (range 0-100) is reported for the BASC-2 assessment. Higher scores reflect greater behavioral problems.
Time Frame: Pretherapy, Week 4, Week 24, End of Therapy, and 6 Months Post End of Therapy
Population: This QOL analysis included patients only within Stratum A.
Measure: Mean (Standard Deviation); unit: T score
Groups:
- Pretherapy: Psychological assessment completed before start of therapy.
- Week 4: Psychological assessment completed at Week 4
- Week 24: Psychological assessment completed at Week 24
Arm/Group | Pretherapy | Week 4 | Week 24 | End of Therapy | 6 Months After End of Therapy
Number analyzed (Participants) | 21 | 21 | 19 | 18 | 16
T score | 44.9 (8.1) | 45.9 (8.3) | 44.2 (6.9) | 47.2 (11.1) | 42.3 (7.2)

23. Other Pre Specified Outcome: BASC-2 Psychological Assessment (Stratum B)
Description: as for outcome 22
Time Frame: Pretherapy, Week 4, Week 24, End of Therapy, and 6 Months Post End of Therapy
Population: Only one patient had evaluable data in Stratum B, but scores were not available for this instrument due to the age of the patient.
Arm/Group | Pretherapy | Week 4 | Week 24 | End of Therapy | 6 Months After End of Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

24. Other Pre Specified Outcome: BRIEF Psychological Assessment (Stratum A)
Description: The Behavioral Rating Inventory of Executive Function (BRIEF) was administered to parents, assessing for any effects on behavior or mood in children undergoing study therapy. The global executive composite (GEC) T-score (range 0-100) is reported for the BRIEF assessment. Higher scores reflect poorer executive function.
Time Frame: Pretherapy, Week 4, Week 24, End of Therapy, and 6 Months Post End of Therapy
Population: This QOL analysis included patients only within Stratum A.
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Pretherapy | Week 4 | Week 24 | End of Therapy | 6 Months After End of Therapy
Number analyzed (Participants) | 17 | 17 | 13 | 14 | 11
T score | 47.9 (12.8) | 50.8 (11.9) | 48.6 (12.4) | 47.6 (12.6) | 42.6 (8.1)

25. Other Pre Specified Outcome: BRIEF Psychological Assessment (Stratum B)
Description: as for outcome 24
Time Frame: Pretherapy, Week 4, Week 24, End of Therapy, and 6 Months Post End of Therapy
Population: as for outcome 23
Arm/Group | Pretherapy | Week 4 | Week 24 | End of Therapy | 6 Months After End of Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events are reported from the start of treatment for the first patient in May 2008 through April 2016.
Arm/Group | Peginterferon ɑ-2b/Non-pegylated Interferon ɑ-2b | Temozolomide/Peginterferon ɑ-2b With Measureable Disease | Temozolomide/Peginterferon ɑ-2b Without Measureable Disease
Serious Adverse Events (participants affected / at risk) | 3/23 | 0/2 | 0/4
Other Adverse Events (participants affected / at risk) | 23/23 | 2/2 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peginterferon ɑ-2b/Non-pegylated Interferon ɑ-2b (N=23) | Temozolomide/Peginterferon ɑ-2b With Measureable Disease (N=2) | Temozolomide/Peginterferon ɑ-2b Without Measureable Disease (N=4)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Confusion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Joint function (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Mood alteration, agitation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Psychosis (hallucinations/delusions) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peginterferon ɑ-2b/Non-pegylated Interferon ɑ-2b (N=23) | Temozolomide/Peginterferon ɑ-2b With Measureable Disease (N=2) | Temozolomide/Peginterferon ɑ-2b Without Measureable Disease (N=4)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 11 (19) | 0 (0) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 13 (29) | 2 (2) | 2 (11)
Leukocytes) total WBC) (Blood and lymphatic system disorders) | 22 (116) | 2 (4) | 4 (16)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 23 (142) | 0 (0) | 4 (16)
Platelets (Blood and lymphatic system disorders) | 15 (28) | 0 (0) | 3 (18)
Supraventricular and nodal arrhythmia, sinus bradycardia (Cardiac disorders) | 8 (20) | 0 (0) | 1 (3)
Supraventricular and nodal arrhythmia, sinus tachycardia (Cardiac disorders) | 9 (22) | 2 (4) | 1 (3)
Hypertension (Cardiac disorders) | 6 (21) | 0 (0) | 2 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 20 (100) | 0 (0) | 3 (4)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC<1.0 x 10e9/L) (General disorders) | 16 (39) | 1 (1) | 2 (3)
Rigors/chills (General disorders) | 10 (19) | 0 (0) | 0 (0)
Sweating (diaphoresis) (General disorders) | 2 (5) | 0 (0) | 0 (0)
Weight gain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Weight loss (General disorders) | 4 (9) | 1 (2) | 1 (1)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 4 (9) | 0 (0) | 0 (0)
Dermatology/skin - other (Skin and subcutaneous tissue disorders) | 4 (7) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0) | 0 (0)
Flushing (Skin and subcutaneous tissue disorders) | 3 (7) | 0 (0) | 1 (1)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 7 (8) | 0 (0) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 20 (83) | 1 (2) | 3 (5)
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hot flashes/flushes (Endocrine disorders) | 3 (3) | 0 (0) | 0 (0)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 3 (5) | 0 (0) | 0 (0)
Anorexia (Gastrointestinal disorders) | 18 (42) | 2 (2) | 2 (3)
Constipation (Gastrointestinal disorders) | 9 (18) | 0 (0) | 0 (0)
Dehydration (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 13 (32) | 1 (1) | 4 (9)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Heartburn/dyspepsia (Gastrointestinal disorders) | 2 (3) | 0 (0) | 1 (1)
Mucositis/stomatitis (clinical exam), oral cavity (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 17 (38) | 0 (0) | 4 (9)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 12 (30) | 0 (0) | 3 (17)
Hemorrhage, GI, lower GI NOS (Vascular disorders) | 3 (4) | 0 (0) | 0 (0)
Hemorrhage, GI, oral cavity (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Hemorrhage, GI, rectum (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Hemorrhage, GI, upper GI NOS (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
Hemorrhage, pulmonary/upper respiratory, nose (Vascular disorders) | 3 (7) | 0 (0) | 0 (0)
Hemorrhage/bleeding - other (Vascular disorders) | 2 (3) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils, lip/perioral (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils, middle ear (otitis media) (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils, nerve-peripheral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils, sinus (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils, upper airway NOS (Infections and infestations) | 3 (4) | 0 (0) | 1 (1)
Infection with unknown ANC, sinus (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Edema: head and neck (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Edema: limb (Blood and lymphatic system disorders) | 2 (5) | 0 (0) | 1 (1)
Edema: trunk/genital (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0)
Lymphatics - other (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (2)
ALT, SGPT (serum gluatmic pyruvic transaminase) (Metabolism and nutrition disorders) | 22 (90) | 0 (0) | 2 (10)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 23 (73) | 1 (1) | 1 (3)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 6 (6) | 1 (1) | 1 (1)
Alkaline phosphatase (Metabolism and nutrition disorders) | 4 (6) | 0 (0) | 0 (0)
Amylase (Metabolism and nutrition disorders) | 8 (14) | 0 (0) | 1 (4)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Calcium, serum-low (hypocalcemia (Metabolism and nutrition disorders) | 3 (5) | 0 (0) | 0 (0)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 12 (23) | 1 (1) | 2 (5)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 10 (14) | 0 (0) | 1 (3)
Lipase (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 2 (5)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 6 (9) | 0 (0) | 0 (0)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 3 (8) | 0 (0) | 0 (0)
Metabolic/laboratory - other (Metabolism and nutrition disorders) | 7 (23) | 0 (0) | 0 (0)
Potassium, serum-high (hyperkalemia (Metabolism and nutrition disorders) | 5 (9) | 0 (0) | 2 (8)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 2 (2)
Proteinuria (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 9 (17) | 0 (0) | 2 (2)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 11 (17) | 0 (0) | 1 (1)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 7 (7) | 0 (0) | 3 (9)
Dizziness (Nervous system disorders) | 3 (5) | 0 (0) | 0 (0)
Mood alteration, agitation (Nervous system disorders) | 9 (23) | 0 (0) | 0 (0)
Mood alteration, anxiety (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1)
Mood alteration, depression (Nervous system disorders) | 3 (4) | 0 (0) | 0 (0)
Neuropathy: sensory (Nervous system disorders) | 5 (8) | 0 (0) | 0 (0)
Personality/behavioral (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Ocular surface disease (Eye disorders) | 2 (3) | 0 (0) | 0 (0)
Ocular/visual - other (Eye disorders) | 2 (3) | 0 (0) | 0 (0)
Vision-blurred vision (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 0 (0) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Incontinence, urinary (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (2)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (2)
Irregular menses (change from baseline) (Reproductive system and breast disorders) | 2 (3) | 0 (0) | 0 (0)
Pain, abdomen NOS (General disorders) | 8 (16) | 1 (2) | 2 (5)
Pain, back (General disorders) | 3 (22) | 1 (1) | 2 (2)
Pain, chest wall (General disorders) | 2 (2) | 0 (0) | 1 (4)
Pain, chest/thorax NOS (General disorders) | 3 (5) | 0 (0) | 2 (3)
Pain, dental/teeth/peridontal (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pain, external ear (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pain, extremity-limb (General disorders) | 12 (27) | 1 (1) | 0 (0)
Pain, head/headache (General disorders) | 18 (257) | 1 (2) | 2 (6)
Pain, joint (General disorders) | 3 (4) | 0 (0) | 0 (0)
Pain, muscle (General disorders) | 6 (12) | 0 (0) | 1 (1)
Pain, neck (General disorders) | 3 (3) | 0 (0) | 0 (0)
Pain, pain NOS (General disorders) | 8 (43) | 0 (0) | 0 (0)
Pain, stomach (General disorders) | 3 (3) | 0 (0) | 0 (0)
Pain, throat/pharynx/larynx (General disorders) | 7 (9) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils, Lung (pnemonia) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 2 (6) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study closed early due to poor accrual to stratum B1.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes